CLINICAL TRIAL: NCT07382063
Title: Effects of Extra-fascial Interscalene Brachial Plexus Block on Diaphragmatic Function in School-Aged Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Jiaqi Shan, anesthesiologist, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-204-(1)
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Diaphragm Movement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra-fascial interscalene brachial plexus block (ISB) (Placebo Comparator)
  Interventions: Procedure: intra-fascial interscalene brachial plexus block (ISB)
- extra-fascial interscalene brachial plexus block (ISB) (Experimental)
  Interventions: Procedure: extra-fascial interscalene brachial plexus block (ISB)

INTERVENTIONS:
Procedure: extra-fascial interscalene brachial plexus block (ISB) — Perform an extra-fascial interscalene brachial plexus block, positioning the needle tip 2-4 mm lateral to the brachial plexus sheath, at a level equidistant between the C5 and C6 roots, measured using the on-screen caliper tool. Inject 0.5 ml/kg of 0.2% ropivacaine for nerve blockade.
  Arms: extra-fascial interscalene brachial plexus block (ISB)
Procedure: intra-fascial interscalene brachial plexus block (ISB) — Perform an intra-fascial interscalene brachial plexus block by penetrating the brachial plexus fascia and injecting 0.5 ml/kg of 0.2% ropivacaine.
  Arms: intra-fascial interscalene brachial plexus block (ISB)

SUMMARY:
The traditional intra-fascial interscalene brachial plexus block (ISB) is already one of the routine anesthesia methods for pediatric upper limb surgeries in clinical practice. This study aims to clarify the effect of the extra-fascial interscalene brachial plexus block on the diaphragm function of school-age children, as well as its analgesic effect, and to compare it with the traditional intra-fascial ISB. It intends to explore a more effective and safer ISB method for children. With the aim of optimizing techniques and accurately evaluating, to balance the benefits of analgesia and safety, and thereby promoting the development of precise pediatric anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age range: School-aged children (6-12 years old).
* Type of surgery: Upper limb surgery.
* ASA classification: Grades I-II.

Exclusion Criteria:

* Infection, anatomical deformity, or tumor at the puncture site.
* Coagulation disorders (INR > 1.4, platelet count < 100 × 10⁹/L).
* History of allergy to local anesthetics (ropivacaine).
* Severe cardiopulmonary or neurological diseases (e.g., epilepsy, myopathy).
* Pre-existing ipsilateral phrenic nerve paralysis or Horner syndrome.
* Preoperative long-term use of analgesics (which may affect efficacy assessment).
* Parent or child refusal to participate in the study.
* Emergency surgery or inability to cooperate with assessments (e.g., severe developmental delay).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the rate of diaphragmatic paralysis using ultrasound. | From enrollment to the end of treatment at 2-3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided